CLINICAL TRIAL: NCT03529435
Title: Project Remission: Maximizing Outcomes With Intensive Treatments for Combat-Related Posttraumatic Stress Disorder
Brief Title: Project Remission: Maximizing Outcomes With Intensive Treatments for Combat-Related PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); South Texas Veterans Health Care System (U.S. Federal Agency); C.R.Darnall Army Medical Center (U.S. Federal Agency); Central Texas Veterans Health Care System (Other); VISN 17 Center of Excellence (U.S. Federal Agency); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-13-2-0065
Record Dates: First submitted 2018-04-13; First posted 2018-05-18 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic Stress Disorder; PTSD; Post-Traumatic Stress; Trauma and Stressor Related Disorders; Trauma; Combat; Military; Veterans; Prolonged Exposure; Exposure Therapy; Behavior Therapy; Psychological Treatment; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators, who are blind to treatment condition, conduct semi-structured interviews to assess PTSD diagnosis at the posttreatment, three-month, and six-month follow-up assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massed Prolonged Exposure (Active Comparator): Participants will complete fifteen weekday 90-minute Prolonged Exposure therapy sessions over three consecutive weeks. If necessary, the treatment window may be extended for another week.
  Interventions: Behavioral: Massed Prolonged Exposure
- Intensive Outpatient Prolonged Exposure (Experimental): The IOP-PE will include the same primary treatment components as the Massed-PE protocol (fifteen weekday 90-minute PE sessions delivered five days a week over a three-week period) plus eight augmentations designed to maximize treatment outcomes. Similar to the Mass-PE, participants will have three consecutive weeks to complete treatment; however, the treatment window may be extended another week if necessary.
  Interventions: Behavioral: Intensive Outpatient Prolonged Exposure

INTERVENTIONS:
Behavioral: Massed Prolonged Exposure — Participants will complete fifteen weekday 90-minute Prolonged Exposure therapy sessions over three consecutive weeks. If necessary, the treatment window may be extended for another week.
  Arms: Massed Prolonged Exposure
Behavioral: Intensive Outpatient Prolonged Exposure — The IOP-PE will include the same primary treatment components as the Massed-PE protocol (fifteen weekday 90-minute PE sessions delivered five days a week over a three-week period) plus eight augmentations designed to maximize treatment outcomes. Similar to the Mass-PE, participants will have three consecutive weeks to complete treatment; however, the treatment window may be extended another week if necessary.
  Arms: Intensive Outpatient Prolonged Exposure

SUMMARY:
The study compares two intensive outpatient behavioral programs (Massed Prolonged Exposure versus Intensive Outpatient Prolonged Exposure) for the treatment of posttraumatic stress disorder (PTSD) in post-9/11 active duty service members and veterans. The researchers hope to learn if these programs improve treatment outcomes. The researchers predict that Intensive Outpatient Prolonged Exposure (IOP-PE) will be better at treating PTSD than Massed-Prolonged Exposure (Massed PE).

DETAILED DESCRIPTION:
With an estimated 200,000 - 600,000 post-9/11 service members and veterans suffering from combat-related posttraumatic stress disorder (PTSD; 7-20% of the 3 million who have deployed), there is an urgent need for accessible therapies that are highly effective in quickly treating PTSD to remission, enabling service members to stay fit for active duty and veterans to integrate well into civilian life. While combat-related PTSD can be successfully treated in post-9/11 active duty service members and veterans, recent studies indicate that they do not derive the same degree of benefit from evidence-based behavioral treatments (e.g., Prolonged Exposure; Cognitive Processing Therapy) as their civilian counterparts. This suggests that combat-related PTSD is uniquely different from PTSD in civilians and that treatments are needed that expand and augment established evidence-based treatments in order to address the distinctive elements of combat-related traumas.

Prolonged Exposure (PE) is the PTSD treatment most extensively evaluated in clinical trials with civilians and veterans, and there is strong scientific evidence to support its efficacy. In standard outpatient PE, patients participate in weekly session over the course of two to three months. However, given military work requirements, participation in standard outpatient services is not always feasible. In the largest PE study with post-911 active duty service members to date conducted by Foa and colleagues in 2018 found PE delivered in a massed format (i.e., ten 90-minute PE sessions delivered on weekdays over 2 weeks) results in similar treatment outcomes to those of PE delivered in the standard spaced format (i.e., ten 90-minute PE sessions delivered over 8 weeks).

The current study expands and augments the previous treatment protocol. More specifically, this study examines whether intensive PE protocols can improve on treatment outcomes for post-9/11 service members and veterans with combat-related PTSD. The purpose of this randomized clinical trial is to compare the efficacy Massed-Prolonged Exposure (Massed-PE, 15 90-minute sessions delivered over three weeks) versus Intensive Outpatient Prolonged Exposure protocol (IOP-PE, 15 days of treatment delivered over three weeks). In comparison with the Massed PE examined by Foa, Massed-PE in this study has been modified to include 50% more sessions and release from duty. IOP-PE has been further augmented and includes the following modifications: (1) the use of a team-based treatment approach; (2) clinic-based completion of daily homework assignments; (3) brief therapist feedback sessions after daily homework assignments; (4) enhanced social support; (5) focusing on patients' three most distressing traumas during imaginal exposure; (6) graduated imaginal exposure starting with the least distressing trauma; (7) an optional telescopic, brief, timeline review of all traumatic events that occurred during previous deployments; and (8) the completion of three posttreatment booster sessions. Up to 400 post-9/11 active duty military and veterans will be consented to obtain data from 230 for analysis. The main outcomes of the study include PTSD diagnoses and symptom severity as measured by the Clinician Administered PTSD Scale for the (CAPS-5) and the PTSD Checklist-for the Diagnostic and Statistical Manual for Mental Disorders, 5th Edition(PCL-5). Participants will be assessed at baseline, while in-treatment and at one-, three-, and six-months after treatment completion. The researchers predict that IOP-PE will result in larger reductions than the Massed-PE in PTSD symptoms at the three follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty military service member or veteran (age 18- 65 years) who deployed in support of combat operations post-9/11 seeking behavioral health treatment for PTSD.
2. PTSD diagnosis as assessed by Clinician-Administered Posttraumatic Stress Scale (CAPS-5).
3. Able to speak and read English (due to standardization of outcome measures)

Exclusion Criteria:

1. Current manic episode or a psychotic symptoms requiring immediate stabilization or hospitalization (as determined by the bipolar and psychosis modules of the MINI).
2. Current and severe alcohol use warranting immediate intervention based on clinical judgment.
3. Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires).
4. Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index-Suicidality Subscale and corroborated by a clinical risk assessment by a credentialed provider)
5. Other psychiatric disorders severe enough to warrant designation as the primary disorder as determined by clinician judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | Baseline to 4 Weeks (Posttreatment)
  Change in scale measurements by the Clinician Administered PTSD Scale (CAPS-5). The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms.Total Score (Range 0-80 with higher scores representing more PTSD symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Peterson, PhD, Principal Investigator — University of Texas Health Science Center at San Antonio; South Texas Veterans Health Care System
Locations (4):
- United States (4):
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Central Texas Veterans Health Care System, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foa EB, McLean CP, Zang Y, Rosenfield D, Yadin E, Yarvis JS, Mintz J, Young-McCaughan S, Borah EV, Dondanville KA, Fina BA, Hall-Clark BN, Lichner T, Litz BT, Roache J, Wright EC, Peterson AL; STRONG STAR Consortium. Effect of Prolonged Exposure Therapy Delivered Over 2 Weeks vs 8 Weeks vs Present-Centered Therapy on PTSD Symptom Severity in Military Personnel: A Randomized Clinical Trial. JAMA. 2018 Jan 23;319(4):354-364. doi: 10.1001/jama.2017.21242. PMID 29362795
- [Background] Cigrang JA, Rauch SA, Mintz J, Brundige AR, Mitchell JA, Najera E, Litz BT, Young-McCaughan S, Roache JD, Hembree EA, Goodie JL, Sonnek SM, Peterson AL; STRONG STAR Consortium. Moving effective treatment for posttraumatic stress disorder to primary care: A randomized controlled trial with active duty military. Fam Syst Health. 2017 Dec;35(4):450-462. doi: 10.1037/fsh0000315. PMID 29283612
- [Background] Cigrang JA, Rauch SA, Mintz J, Brundige A, Avila LL, Bryan CJ, Goodie JL, Peterson AL; STRONG STAR Consortium. Treatment of active duty military with PTSD in primary care: A follow-up report. J Anxiety Disord. 2015 Dec;36:110-4. doi: 10.1016/j.janxdis.2015.10.003. Epub 2015 Oct 22. PMID 26519833
- [Background] Steenkamp MM, Litz BT, Hoge CW, Marmar CR. Psychotherapy for Military-Related PTSD: A Review of Randomized Clinical Trials. JAMA. 2015 Aug 4;314(5):489-500. doi: 10.1001/jama.2015.8370. PMID 26241600
- [Background] Blount TH, Cigrang JA, Foa EB, Ford HL, Peterson, AL. Intensive outpatient prolonged exposure for combat-related PTSD: A case study. Cognitive and Behavioral Practice. 2014; 21, 89-96. doi:10.1016/j.cbpra.2013.05.004
- [Background] Foa EB, Hembree EA, Rothbaum, BO. Prolonged exposure therapy for PTSD: Emotional processing of traumatic experiences therapist guide. New York, NY: Oxford University Press. 2007.
- [Background] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Background] Resick PA, Wachen JS, Mintz J, Young-McCaughan S, Roache JD, Borah AM, Borah EV, Dondanville KA, Hembree EA, Litz BT, Peterson AL. A randomized clinical trial of group cognitive processing therapy compared with group present-centered therapy for PTSD among active duty military personnel. J Consult Clin Psychol. 2015 Dec;83(6):1058-1068. doi: 10.1037/ccp0000016. Epub 2015 May 4. PMID 25939018
- [Background] Bisson JI, Ehlers A, Matthews R, Pilling S, Richards D, Turner S. Psychological treatments for chronic post-traumatic stress disorder. Systematic review and meta-analysis. Br J Psychiatry. 2007 Feb;190:97-104. doi: 10.1192/bjp.bp.106.021402. PMID 17267924
- [Background] Peterson AL, Foa EB, Riggs DS. Prolonged exposure therapy for combat-related PTSD. In B. A. Moore, & W. Penk (Eds.), Treating PTSD in military personnel: A clinical handbook (pp. 42-58). New York, NY: Guilford. 2011.
- [Background] Peterson AL, Luethcke CA, Borah EV, Borah AM, Young-McCaughan S. Assessment and treatment of combat-related PTSD in returning war veterans. J Clin Psychol Med Settings. 2011 Jun;18(2):164-75. doi: 10.1007/s10880-011-9238-3. PMID 21626355
- [Background] Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clin Psychol Rev. 2010 Aug;30(6):635-41. doi: 10.1016/j.cpr.2010.04.007. Epub 2010 May 2. PMID 20546985
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.). Washington, DC: Author. 2013.
- [Background] Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr, PP. The PTSD Checklist for DSM-5 (PCL-5). Instrument available from the National Center for PTSD at www.ptsd.va.gov. 2013.
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Derived] Peterson AL, Blount TH, Foa EB, Brown LA, McLean CP, Mintz J, Schobitz RP, DeBeer BR, Mignogna J, Fina BA, Evans WR, Synett S, Hall-Clark BN, Rentz TO, Schrader C, Yarvis JS, Dondanville KA, Hansen H, Jacoby VM, Lara-Ruiz J, Straud CL, Hale WJ, Shah D, Koch LM, Gerwell KM, Young-McCaughan S, Litz BT, Meyer EC, Blankenship AE, Williamson DE, Roache JD, Javors MA, Sharrieff AM, Niles BL, Keane TM; Consortium to Alleviate PTSD. Massed vs Intensive Outpatient Prolonged Exposure for Combat-Related Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2249422. doi: 10.1001/jamanetworkopen.2022.49422. PMID 36602803
- See also: STRONG STAR-CAP website — http://www.strongstar.org